CLINICAL TRIAL: NCT01188668
Title: An Open-Label, 2-Period Sequential Drug Interaction Study To Evaluate The Effect Of A 100 Mg Dose Of Desvenlafaxine SR On The Pharmacokinetics Of Aripiprazole When Coadministered In Healthy Subjects
Brief Title: Open Label Drug Interaction Study Evaluating Desvenlafaxine Succinate Sustained Release (DVS SR) 100mg On The Pharmacokinetics Of Aripiprazole When Coadministered To Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B2061026; 3151A1-1207
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Pharmacokinetics; Cytochrome P-450 CYP2D6; CYP3A4 Protein, Human
Keywords: Pharmacokinetic; safety and tolerability; genetic testing; CYP 2D6 and CYP 3A4
MeSH Terms: interventions — Aripiprazole; Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole + Desvenlafaxine SR (Experimental)
  Interventions: Drug: Aripiprazole; Drug: Aripiprazole + desvenlafaxine succinate sustained release

INTERVENTIONS:
Drug: Aripiprazole — Period 1-Aripiprazole 5mg on study day 1.
  Other Names: DVS-233; Pristiq
Drug: Aripiprazole + desvenlafaxine succinate sustained release — Period 2-Desvenlafaxine SR 100mg on days 1-19 with coadministration of Aripiprazole 5mg on day 7.

SUMMARY:
The goal of this study is to evaluate the effect of multiple doses of Desvenlafaxine Sustained Release (SR) on the pharmacokinetics of Aripiprazole when coadministered to healthy adult subjects. This study will also evaluate the safety and tolerability of Desvenlafaxine SR and Aripiprazole when coadministered to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2 and a total body weight >50 kg (110 lbs)
* Nonsmoker or smoker of fewer than 5 cigarettes per day as determined by history
* An informed consent document signed and dated by the subject

Exclusion Criteria:

* History of significant blood, kidney, endocrine, lung, gastrointestinal, heart, liver, psychiatric, neurologic, or allergic disease
* History of seizure disorder
* Presence or history of glaucoma or increased intraocular pressure
* Allergy to or unable to tolerate aripiprazole, desvenlafaxine, or venlafaxine
* History of substance abuse within 1 year of study
* A positive urine drug screen
* Treatment with an investigational drug within 30 days
* Consumption of grapefruit or grapefruit related citrus fruits
* 12 lead ECG demonstrating QTc >450 msec at screening
* Pregnant or nursing females
* Use of prescription or nonprescription drugs and dietary supplements
* History of sensitivity to heparin or heparin induced thrombocytopenia
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole 5 mg, Aripiprazole 5 mg + DVS SR 100 mg: Aripiprazole (ARIP) as a single oral dose of 5 milligrams (mg) Period 1 / Day 1. Desvenlafaxine sustained release (DVS SR) as a single oral dose of 100 mg Period 2 / Day 1 through Day 6 (steady state) and Day 7 though 19. Aripiprazole as a single oral dose of 5 mg coadministered with the DVS SR dose on Period 2 / Day 7.
Period: Period 1: ARIP Alone
Arm/Group | Aripiprazole 5 mg, Aripiprazole 5 mg + DVS SR 100 mg
Started | 38
Completed | 36
Not Completed | 2
Not completed — Protocol Violation | 2
Period: Period 2: Coadministration ARIP + DVS SR
Arm/Group | Aripiprazole 5 mg, Aripiprazole 5 mg + DVS SR 100 mg
Started | 36
Completed | 33
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole 5 mg, Aripiprazole 5 mg + DVS SR 100 mg: Aripiprazole as a single oral dose of 5 mg Period 1 / Day 1. DVS SR as a single oral dose of 100 mg Period 2 / Day 1 through Day 6 (steady state) and Day 7 though 19. Aripiprazole as a single oral dose of 5 mg coadministered with the DVS SR dose on Period 2 / Day 7.
Arm/Group | Aripiprazole 5 mg, Aripiprazole 5 mg + DVS SR 100 mg
Number analyzed (Participants) | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 35.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Aripiprazole Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞); measured as nanograms multiplied by hours divided by milliliters (ng*hr/mL).
Time Frame: Period 1 / Day 1: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 120, 168, 216, 264, and 312 hours after dosing; Period 2 / Day 7: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours after dosing; also 0 hour Period 2 / Day 8, 9, 10, 12, 14, 16, 18, and Day 20
Population: Pharmacokinetic (PK) parameter analysis population: all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. N=Number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Aripiprazole 5 mg (Period 1): Aripiprazole as a single oral dose of 5 mg Period 1 / Day 1.
- Aripiprazole 5 mg + DVS SR 100 mg (Period 2): DVS SR as a single oral dose of 100 mg Period 2 / Day 1 through Day 6 (steady state) and Day 7 though 19. Aripiprazole as a single oral dose of 5 mg coadministered with the DVS SR dose on Period 2 / Day 7.
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 37 | 35
ng*hr/mL | 1494 (699.98) | 1604 (561.45)
Statistical Analysis 1: Comparison: Aripiprazole 5 mg (Period 1) vs Aripiprazole 5 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Aripiprazole 5 mg (test) versus Aripiprazole 5 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 105.97, 90% CI 2-sided [101.39 to 110.76] — Values have been back-transformed from the log scale

2. Secondary Outcome: Aripiprazole Maximum Observed Plasma Concentration (Cmax) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Cmax measured as nanograms per milliliters (ng/mL).
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=Number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 38 | 35
ng/mL | 24.66 (7.6031) | 24.69 (7.4186)
Statistical Analysis 1: Comparison: Aripiprazole 5 mg (Period 1) vs Aripiprazole 5 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Aripiprazole 5 mg (test) versus Aripiprazole 5 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 101.05, 90% CI 2-sided [92.94 to 109.87] — Values have been back-transformed from the log scale

3. Secondary Outcome: Aripiprazole Time for Cmax (Tmax) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Time for maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=Number of participants contributing to the median.
Measure: Median (Full Range); unit: hours
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 38 | 35
hours | 3.00 [2.00 to 8.00] | 4.00 [2.00 to 8.00]

4. Secondary Outcome: Aripiprazole Terminal Half-life (t 1/2) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=Number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 38 | 35
hours | 85.17 (22.191) | 84.18 (20.025)

5. Secondary Outcome: Aripiprazole Apparent Clearance (CL/F) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood calculated as (Dose/AUCinf); measured as milliliters per minute (mL/min).
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=Number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: mL/min
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 37 | 35
mL/min | 55.76 (25.345) | 51.92 (19.655)

6. Secondary Outcome: Aripiprazole Apparent Volume of Distribution (Vz/F) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Calculated as Dose / (AUCinf * kel); where kel=terminal phase rate constant.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=Number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: liters
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 37 | 35
liters | 397.3 (129.28) | 368.1 (102.01)

7. Secondary Outcome: Dehydro-aripiprazole (Metabolite) Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Dehydro-aripiprazole is a metabolite of Aripiprazole. Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=Number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 18 | 14
ng*hr/mL | 695.9 (151.95) | 685.8 (148.14)
Statistical Analysis 1: Comparison: Aripiprazole 5 mg (Period 1) vs Aripiprazole 5 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Aripiprazole 5 mg (test) versus Aripiprazole 5 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 102.93, 90% CI 2-sided [94.21 to 112.46] — Values have been back-transformed from the log scale

8. Secondary Outcome: Dehydro-aripiprazole (Metabolite) Maximum Observed Plasma Concentration (Cmax) Following Aripiprazole Alone and When Coadministered With DVS SR
Time Frame: Period 1 / Day 1: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 120, 168, 216, 264, and 312 hours after dosing; Period 2 / Day 7: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours after dosing
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 38 | 35
ng/mL | 3.007 (1.0889) | 3.185 (1.0127)
Statistical Analysis 1: Comparison: Aripiprazole 5 mg (Period 1) vs Aripiprazole 5 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Aripiprazole 5 mg (test) versus Aripiprazole 5 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 106.27, 90% CI 2-sided [100.97 to 111.85] — Values have been back-transformed from the log scale

9. Secondary Outcome: Dehydro-aripiprazole (Metabolite) Time for Cmax (Tmax) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Time for maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Median (Full Range); unit: hours
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 38 | 35
hours | 59.9 [23.9 to 120] | 71.9 [23.9 to 168]

10. Secondary Outcome: Dehydro-aripiprazole (Metabolite) Terminal Half-life (t 1/2) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=Number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 18 | 14
hours | 97.78 (16.588) | 94.27 (16.403)

11. Secondary Outcome: Dehydro-aripiprazole (Metabolite) Apparent Clearance (CL/F) Following Aripiprazole Alone and When Coadministered With DVS SR
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood calculated as (Dose/AUCinf).
Time Frame: as for outcome 1
Population: PK parameter analysis population. Data was insufficient for analysis; not analyzable.
Measure: Geometric Mean (Standard Deviation); unit: mL/min
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Dehydro-aripiprazole (Metabolite) Apparent Volume of Distribution (Vz/F) Following Aripiprazole Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population. Data was insufficient for analysis; not analyzable.
Measure: Geometric Mean (Standard Deviation); unit: liters
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Plasma Aripiprazole Concentration Versus Time Summary: Aripiprazole 5mg, DVS SR 100 mg + Aripiprazole 5 mg
Description: Summary statistics were to be calculated by setting concentration values below the lower limit of quantification (LLQ = 0.100 ng/mL) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) = 0.
Time Frame: Period 1 / Day 1 and Period 2 / Day 1: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 120, 168, 216, 264, and 312 hours after dosing
Population: PK concentration analysis population: all randomized and treated participants who had at least 1 concentration in at least 1 treatment period. Period 2 / Day 1 = Day 1 of Aripiprazole dosing (Period 2 / Day 7) within the DVS SR, Aripiprazole coadministration dosing period.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 38 | 35
ng/mL
  0 hour | NA [NA to NA] — No observations above the lower limit of quantification. | 0.1290 [0.000 to 0.813]
  0.5 hour post dose | 0.4800 [0.000 to 6.65] | 1.220 [0.000 to 7.57]
  1 hour post dose | 10.69 [0.000 to 26.9] | 9.545 [0.167 to 33.1]
  2 hours post dose | 23.40 [1.07 to 46.7] | 21.70 [0.824 to 44.1]
  3 hours post dose | 21.75 [3.01 to 37.2] | 24.40 [8.27 to 36.1]
  4 hours post dose | 21.35 [5.59 to 35.1] | 25.40 [8.85 to 31.9]
  6 hours post dose | 18.95 [9.96 to 27.9] | 20.70 [7.22 to 25.8]
  8 hours post dose | 16.65 [8.39 to 23.7] | 18.00 [7.24 to 23.8]
  12 hours post dose | 13.65 [6.53 to 23.7] | 13.80 [6.46 to 19.2]
  16 hours post dose | 11.50 [5.73 to 18.2] | 12.50 [5.84 to 18.7]
  24 hours post dose | 10.70 [5.35 to 18.1] | 12.20 [5.47 to 18.6]
  48 hours post dose | 8.310 [3.88 to 14.2] | 8.940 [4.64 to 13.5]
  72 hours post dose | 6.255 [2.46 to 11.6] | 6.870 [3.36 to 11.1]
  120 hours post dose | 3.680 [1.63 to 10.1] | 4.000 [1.88 to 7.82]
  168 hours post dose | 2.390 [0.926 to 16.3] | 2.720 [0.872 to 5.53]
  216 hours post dose | 1.730 [0.491 to 13.4] | 1.960 [0.457 to 4.30]
  264 hours post dose | 1.080 [0.337 to 4.41] | 1.340 [0.237 to 3.20]
  312 hours post dose | 0.8040 [0.202 to 3.99] | 1.010 [0.128 to 2.58]

14. Secondary Outcome: Plasma Dehydro-aripiprazole (Metabolite) Concentration Versus Time Summary: Aripiprazole 5mg, DVS SR 100 mg, Aripiprazole 5 mg
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Aripiprazole 5 mg (Period 1) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 38 | 35
ng/mL
  0 hour | NA [NA to NA] — No observations above the lower limit of quantification. | 0.1640 [0.000 to 0.871]
  0.5 hour post dose | 0.0000 [0.0000 to 0.138] | 0.2120 [0.000 to 0.950]
  1 hour post dose | 0.2740 [0.000 to 1.38] | 0.5965 [0.000 to 1.64]
  2 hours post dose | 0.9470 [0.000 to 4.29] | 1.240 [0.132 to 2.64]
  3 hours post dose | 1.260 [0.115 to 5.55] | 1.660 [0.473 to 3.33]
  4 hours post dose | 1.495 [0.277 to 5.38] | 1.880 [0.791 to 4.13]
  6 hours post dose | 1.650 [0.453 to 5.57] | 1.910 [0.686 to 4.72]
  8 hours post dose | 1.780 [0.689 to 5.80] | 1.910 [0.686 to 5.29]
  12 hours post dose | 1.845 [0.748 to 5.35] | 1.950 [0.654 to 5.15]
  16 hours post dose | 2.010 [0.819 to 5.16] | 1.970 [0.695 to 4.77]
  24 hours post dose | 2.520 [1.01 to 6.29] | 2.550 [0.952 to 5.68]
  48 hours post dose | 3.135 [1.26 to 5.79] | 3.160 [1.00 to 5.43]
  72 hours post dose | 2.935 [1.31 to 4.61] | 3.020 [1.06 to 6.08]
  120 hours post dose | 2.440 [1.25 to 4.16] | 2.360 [1.14 to 4.16]
  168 hours post dose | 1.920 [0.996 to 3.76] | 1.980 [1.09 to 3.43]
  216 hours post dose | 1.570 [0.650 to 3.17] | 1.460 [0.744 to 2.96]
  264 hours post dose | 1.080 [0.429 to 3.13] | 1.130 [0.454 to 2.57]
  312 hours post dose | 0.8660 [0.248 to 2.85] | 0.9680 [0.252 to 2.10]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 27 (follow-up telephone visit)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. Participants are counted for each treatment sequence.
Groups:
- DVS SR 100 mg (Period 2): DVS SR as a single oral dose of 100 mg Period 2 / Day 1 through Day 6 (steady state).
- Aripiprazole 5 mg + DVS SR 100 mg (Period 2): DVS SR as a single oral dose of 100 mg Period 2 / Day 7 though Day 19. Aripiprazole as a single oral dose of 5 mg coadministered with the DVS SR dose on Period 2 / Day 7.
Arm/Group | Aripiprazole 5 mg (Period 1) | DVS SR 100 mg (Period 2) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2)
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 14/38 | 5/36 | 9/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 5 mg (Period 1) (N=38) | DVS SR 100 mg (Period 2) (N=36) | Aripiprazole 5 mg + DVS SR 100 mg (Period 2) (N=35)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 2 | 5
Salivary gland pain (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 2
Presyncope (Nervous system disorders) | 2 | 0 | 1
Attention deficit / hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 7 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.